CLINICAL TRIAL: NCT04822974
Title: TORQUETENOVIRUS IN CAR-T THERAPY: PREDICTION OF THE RISK OF CYTOKINE RELEASE SYNDROME AND DIFFERENTIAL DIAGNOSIS WITH INFECTION
Brief Title: TORQUETENOVIRUS IN CAR-T THERAPY: PREDICTION OF THE CRS
Acronym: TTV-CART
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institut Paoli-Calmettes (Other)
Collaborators: Hospital Clínico Universitario de Valencia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TTV-CART-IPC 2020-063
Record Dates: First submitted 2021-03-24; First posted 2021-03-30 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Hematologic Cancer
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- STUDY ARM (Experimental): blood samples collection
  Interventions: Other: blood collection

INTERVENTIONS:
Other: blood collection — longitudinally collection of blood samples for each patient included.

SUMMARY:
Torque Teno Virus (TTV) prevalence in the general population is very high (>90%) and has not been consistently confirmed to cause any disease. Kidney transplant studies seem to indicate that an elevated viremia could predict the risk of de-veloping an infectious process in the following weeks. An study of the influence of TTV as a predictive marker of infection in kidney transplant recipi-ents showed higher TTV levels, even 3 months before the infectious process, allowing the authors to postulate that the quantification of TTV could help to modulate the treatment of patients at risk. Publications of subsequent studies seem to confirm these data.In the field of hematopoietic stem cell transplantation (HSCT) few studies have analyzed the replication kinetics of TTV. There seems to be a drop in TTV plasma load after conditioning treatment, with a progressive increase in the first months post-transplant, in parallel with the number of lymphocytes. In early stages of HSCT, a relation-ship between TTV replication kinetics and the probability of developing an infection by CMV has also been described. Likewise, the possible relationship of TTV with other complications of HSCT, such as Epstein-Barr virus infection (EBV) or graft-versus-host disease (GvHD), have been reported. However, not every study conducted to date show this line of results.

DETAILED DESCRIPTION:
Torque Teno Virus (TTV) is the prototype of the Anelloviridae family-single chain and circular viruses. These viruses form about 70% of the human virome. TTV prevalence in the general population is very high (>90%) and has not been consistently confirmed to cause any disease. Kidney transplant studies seem to indicate that an elevated viremia could predict the risk of de-veloping an infectious process (bacterial, viral or fungal) in the following weeks. A group of research analyzed the influence of TTV as a predictive marker of infection in 169 kidney transplant recipi-ents. Patients with infection showed higher TTV levels, even 3 months before the infectious process, allowing its authors to postulate that the quantification of TTV could help to modulate the treatment of patients at risk (reducing immunosuppression, introducing or prolonging antimi-crobial prophylaxis). Publications of subsequent studies with greater number of patients seem to confirm these data. Likewise, in the specific case of CMV infection, the quantification of TTV in the early stages of kidney or liver transplantation also allows identification of patients at risk of developing a CMV infection. In the field of hematopoietic stem cell transplantation (HSCT) few studies have analyzed the replication kinetics of TTV. There seems to be a drop in TTV plasma load after conditioning treatment, with a progressive increase in the first months post-transplant, in parallel with the number of lymphocytes. In early stages of HSCT, a relation-ship between TTV replication kinetics and the probability of developing an infection by CMV has also been described. Likewise, the possible relationship of TTV with other complications of HSCT, such as Epstein-Barr virus infection (EBV) or graft-versus-host disease (GvHD), have been reported. However, not every study conducted to date show this line of results. An other research analyzed 2054 blood samples from 123 patients undergoing HSCT, finding no significant differences between TTV and post-transplant complications, such as viral reactivations (CMV, EBV or adenovirus), acute GvHD, relapse or mortality

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (>=18 years).
2. Patient going to be treated by CAR-T Cell therapy
3. Able to comply with the protocol.
4. Written informed consent.
5. Patient affiliated to the national "Social Security" regimen or beneficiary of this regimen

Exclusion Criteria:

1. Pregnancy/breast feeding.
2. Patient considered socially or psychologically unable to comply with the treatment and the required medical follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Plasma viral load and TTV replication kinetics | d0, d1, d3, d5, d7, d10, d14, d21, d28, d60 and d90 after CAR-T Cell treatment
  comparaition between before during and after CART

SECONDARY OUTCOMES:
Plasma viral load and CMV replication kinetics | d0, d14, d28, d60 and d90 after CAR-T Cell treatment
  comparaition between before during and after CART
infections | 100 days
  Reported infections during the study
Cytokines | d0, d3, d7, d10 and d14 after CAR-T Cell treatment
  Cytokines comparison between samples

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Benzaquen A, Gimenez E, Iacoboni G, Guerreiro M, Hernani R, Albert E, Carpio C, Balaguer A, Perez A, S de la Asuncion C, Sanchez-Salinas MA, Chorao P, Pinana JL, Beas F, Montoro J, Hernandez-Boluda JC, Facal A, Ferrer B, Villalba M, Amat P, Gomez MD, Campos D, Terol MJ, Sanz J, Barba P, Navarro D, Solano C. Torque Teno Virus plasma DNA load: a novel prognostic biomarker in CAR-T therapy. Bone Marrow Transplant. 2024 Jan;59(1):93-100. doi: 10.1038/s41409-023-02114-0. Epub 2023 Nov 2. PMID 37919456